CLINICAL TRIAL: NCT05317117
Title: Evaluating the Clinical Performance and Usability of Novel Malaria Rapid Diagnostic Tests (RDTs) for the Detection of Plasmodium Malaria Infections in Brazil
Brief Title: Evaluating the Clinical Performance and Usability of Novel Malaria RDTs in Brazil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PATH (Other)
Collaborators: Centro de Pesquisa em Medicina Tropical de Rondonia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1807405
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2021-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NxTek™ Malaria P.f plus Rapid Diagnostic Test (RDT) and NxTek™ Malaria P.f/P.v RDT (Other): All participants will be tested with two investigational IVDs at the point of care, the NxTek™ Malaria P.f plus Rapid Diagnostic Test (RDT) and the NxTek™ Malaria P.f/P.v RDT, in addition to comparator tests and the standard of care (microscopy). The investigational tests will not be used to determine any treatment or case management.
  Interventions: Diagnostic Test: NxTek™ Malaria P.f plus Rapid Diagnostic Test (RDT) and NxTek™ Malaria P.f/P.v RDT

INTERVENTIONS:
Diagnostic Test: NxTek™ Malaria P.f plus Rapid Diagnostic Test (RDT) and NxTek™ Malaria P.f/P.v RDT — The NxTek (TM) Malaria Pf Plus, developed by Abbott, is a sensitive rapid chromatographic immunoassay for the qualitative detection of histidine-rich protein 2 (HRP2) and pLDH on a single test line of Pf malaria in human whole blood. This test is a lateral flow test for in vitro professional diagnostic use and intended as an aid to early diagnosis of Malaria infection in-patients with clinical symptoms.
  The NxTek (TM) Malaria Pf/Pv Plus, developed by Abbott, is a sensitive rapid chromatographic immunoassay for the qualitative detection of histidine-rich protein 2 (HRP2) and Plasmodium lactate dehydrogenase (pLDH) of Plasmodium falciparum (Pf) on one test line and of pLDH of Plasmodium vivax (Pv) malaria on a second test line in human whole blood. This test is a lateral flow test for in vitro professional diagnostic use and intended as an aid to early diagnosis of Malaria infection in-patients with clinical symptoms.

SUMMARY:
Prospective cross-sectional diagnostic accuracy study with 1,000 patient participants and 30 lay provider/health care worker participants. The patient participant population will be recruited at clinics. At the point of care, study staff will collect capillary blood samples and conduct malaria microscopy (both the standard of care and study specific research-grade microscopy) and two index tests: the NxTek™ Malaria P.f plus Rapid Diagnostic Test (RDT) and the NxTek™ Malaria P.f/P.v RDT. Venous blood will be collected and transferred to the laboratory where the reference PCR assay and three comparator RDTs will be run. The index RDTs will also be repeated in the laboratory. All clinical management of study participants will follow the standard of care for malaria diagnosis in Brazil and will be based on the standard microscopy result. Confirmatory testing may also be conducted, such as typing and sequencing of Plasmodium genes and antigens of interest, including but not limited to HRP2, HRP3, and pLDH as well as the human inflammatory response marker CRP.

The lay provider/health worker participants will include intended users of the index tests. They will be surveyed to assess index test usability through a questionnaire to assess label and packaging comprehension as well as results interpretation.

DETAILED DESCRIPTION:
Primary Objectives

1.1 To assess the sensitivity, specificity and, when applicable, positive and negative predicting values (PPV and NPV) [altogether referred to hereafter as "diagnostic accuracy"] of NxTek™ Malaria Pf Plus in intended use settings for detecting P. falciparum infections in capillary whole blood samples collected prospectively from patients with symptoms suggestive of malaria.

1.2 To assess the diagnostic accuracy of NxTek™ Malaria Pf/Pv Plus in intended use settings for detecting P. falciparum and P. vivax infections in capillary whole blood samples collected prospectively from patients with symptoms suggestive of malaria.

Secondary Objectives

2.1 To assess the diagnostic accuracy of the study comparator tests in intended use settings for detecting P. falciparum and P. vivax infections in venous whole blood samples collected prospectively from patients with symptoms suggestive of malaria.

1.3 To determine the frequency of P. falciparum infections containing HRP2 and/or HRP3 mutations and assess the impact of those on HRP2-based RDT diagnostic accuracy.

1.4 To assess the comprehension of the test packaging and labeling among intended users (trained lay providers and trained health care workers).

1.5 To assess the ability to read and interpret the test result outputs among intended users (trained lay providers and trained health care workers).

ELIGIBILITY:
Inclusion Criteria (diagnostic accuracy):

* Aged 2 years of age or older
* Presenting at the study site with fever or a history of fever during the preceding 48-hours
* Freely agreeing to participate by providing informed consent (and assent, as applicable)

Exclusion Criteria (diagnostic accuracy):

- Presence of symptoms and signs of severe illness and/or central nervous system infections as defined by WHO guidelines

Inclusion Criteria (usability):

* Aged 18 years of age or older
* Provides malaria case management at the study site
* Considered an intended user of the index tests (lay user or healthcare worker)
* Freely agreeing to participate by providing informed consent

Exclusion Criteria (usability):

None

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1030 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of NxTek™ Malaria Pf Plus for the detection of P. falciparum infections | 5 months
  1.1 Estimates of diagnostic accuracy characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV) of NxTek™ Malaria Pf Plus for the detection of P. falciparum infections in patients with symptoms suggestive of malaria.
Diagnostic accuracy of of NxTek™ Malaria Pf/Pv Plus for the detection of P. falciparum and P.vivax infections | 5 months
  1.2 Estimates of diagnostic accuracy characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV) of NxTek™ Malaria Pf/Pv Plus for the detection of P. falciparum and P.vivax infections in patients with symptoms suggestive of malaria.

SECONDARY OUTCOMES:
Diagnostic accuracy of comparator tests for the detection of P. falciparum and, when relevant, P.vivax infections | 5 months
  2.1 Estimates of diagnostic accuracy characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV) of comparator tests for the detection of P. falciparum and, when relevant, P.vivax infections in patients with symptoms suggestive of malaria.
Frequency of P. falciparum infections containing HRP2 and/or HRP3 mutations. | 5 months
  2.2 Frequency of P. falciparum infections containing HRP2 and/or HRP3 mutations.
Diagnostic accuracy of the index tests for the detection of P. falciparum infections with HRP2 and/or HRP3 deletions | 5 months
  2.3 Estimates of diagnostic accuracy characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV) of the index tests for the detection of P. falciparum infections with HRP2 and/or HRP3 deletions in patients with symptoms suggestive of malaria.
Usability: label comprehension | 1 week
  2.4 Percent of end users who can accurately comprehend key messaging included in the investigational device packaging and labels.
Usability: results interpretation | 1 week
  2.5 Percent of end users who can accurately interpret the investigational device result output.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Domingo, PhD, Principal Investigator — PATH
Locations (1):
- Centro de Pesquisa em Medicina Tropical de Rondônia (CEPEM), Porto Velho, Rondônia, Brazil

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any IPD with other researchers.